CLINICAL TRIAL: NCT02149381
Title: Psychosocial Group Interventions for Depression: Systemic and Neurophysiological Correlates of Treatment Effect. A Randomized, Controlled Trial
Brief Title: Psychosocial Group Interventions for Depression
Acronym: PsySysNe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Jyväskylä Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PsySysNe
Record Dates: First submitted 2014-04-07; First posted 2014-05-29 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Depression
Keywords: Depression; treatment as usual; CBASP; befriending
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBASP (Experimental): Cognitive Behavioral System of Psychotherapy is a manual-based group intervention for chr depression (20 weeks).
  Interventions: Behavioral: CBASP; Other: Treatment as usual
- Befriending (Active Comparator): Befriending is a social support intervention
  Interventions: Behavioral: CBASP; Other: Treatment as usual
- Treatment as usual (Active Comparator): Conventional psychiatric outpatient treatment (individual counseling)
  Interventions: Behavioral: CBASP; Behavioral: Befriending

INTERVENTIONS:
Behavioral: CBASP — Cognitive behavioral group intervention for individuals suffering from chronic depression
Behavioral: Befriending — Social support intervention, sessions once per week
  Arms: Treatment as usual
Other: Treatment as usual — Conventional psychiatric outpatient treatment (individual counseling)
  Arms: Befriending; CBASP

SUMMARY:
A total of 384 patients suffering from chronic depressive disorder will be randomized to receive treatment as usual, CBASP, or befriending for a period of five months. The primary outcome is change in Montgomery-Åsberg Depression Scale. Secondary outcomes include changes in self-reported psychiatric symptoms, biomarkers determined from venous blood samples, and neurophysiological parameters. The data gathering is performed at pre- and post intervention stages (i.e., at baseline and at five months). A follow-up questionnaire is sent to the participants six months after the intervention.

DETAILED DESCRIPTION:
The efficacy of 20-week group-CBASP as compared to TAU is evaluated by RCT in a psychiatric outpatient clinics. The recruition is completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Moderate or severe major depression with duration of a minimum of two years OR "double depression" (dysthymia and moderate/severe major depression simultaneously) OR moderate or severe major depression with duration of a minimum of two years, only partially remitted during the time period

Exclusion Criteria:

* Psychotic disorder
* Bipolar disorder
* Current substance abuse (excluding nicotine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Depression | At baseline and after intervention (at 5 months)
  Montgomery-Åsberg Depression Rating Scale

SECONDARY OUTCOMES:
Peripheral blood biomarkers | At baseline and after intervention (at 5 mos)
  Blood samples are collected before and after intervention.

OTHER OUTCOMES:
Neurophysiological measurements. | At baseline and after intervention (5 mos)
  eeg

CONTACTS AND LOCATIONS:
Overall Officials: Soili Lehto, Professor, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Northern Savonia, Finland